CLINICAL TRIAL: NCT03539276
Title: The OptimaMed Intervention to Reduce Inappropriate Medications in Long-term Care Residents With Severe Dementia: Results From a Quasi-experimental Intervention Study
Brief Title: An Intervention to Reduce Inappropriate Medications in Long-term Care Residents With Severe Dementia
Acronym: OptimaMed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: McGill University (Other); Université de Montréal (Other); Université de Sherbrooke (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Dre Edeltraut Kröger, Adjunct professor, CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: OptimaMed-1
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Dementia; Inappropriate Prescribing
Keywords: quality improvement; long term care; polypharmacy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Pre-post study
Who Masked: Participant
Masking Description: It was unlikely that participants could foresee whether or when their medications have been reviewed or modified.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Usual care
- Post-intervention (Experimental): One 90-minute interdisciplinary knowledge exchange including the provision of a validated list of appropriate and inappropriate medications for severe dementia long-term care residents.
  Interventions: Behavioral: Knowledge exchange

INTERVENTIONS:
Behavioral: Knowledge exchange — OptimaMed
  Arms: Post-intervention

SUMMARY:
An education intervention to promote medication reviews and interdisciplinary discussions within long-term care facilities with the aim of improving medication regimen among residents with severe dementia

DETAILED DESCRIPTION:
A quasi-experimental study in three long-term care facilities. The intervention comprises an information leaflet for families of residents, a 90-minute knowledge exchange session for general practitioners, pharmacists and nurses and a list of "generally", "sometimes", and "exceptionally" appropriate medications for severe dementia residents

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia of any etiology
* severe dementia

Exclusion Criteria:

* admission less than 2 months before intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Medication regimen | Four months post intervention
  Active prescriptions

SECONDARY OUTCOMES:
Level of pain | Four months post intervention
  Pain Assessment Checklist for Seniors with Limited Ability to Communicate (PACSLAC).
  The French version of the PACSLAC tool is a validated observational scale in use in Quebec to assess discomfort / pain.
  One point is added to the score for each PACSLAC item (n=60) observed over a 15-minute observation period; the sum of the four 15-minute observation periods gives the total score. The total score ranges from zero to sixty where zero represents no discomfort or pain and sixty a very high level of discomfort or pain.
Level of agitation | Four months post intervention
  Cohen-Mansfield Agitation Inventory () measures level of agitation. Sum of the number of times the Cohen-Mansfield Agitation Inventory items were observed during the four 15-minute observation periods.. The total score ranges from zero to one hundred where zero represents no agitation and one hundred a very high level of agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Edeltraut Kröger, Ph.D., Principal Investigator — Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale
Locations (1):
- Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroger E, Wilchesky M, Marcotte M, Voyer P, Morin M, Champoux N, Monette J, Aubin M, Durand PJ, Verreault R, Arcand M. Medication Use Among Nursing Home Residents With Severe Dementia: Identifying Categories of Appropriateness and Elements of a Successful Intervention. J Am Med Dir Assoc. 2015 Jul 1;16(7):629.e1-17. doi: 10.1016/j.jamda.2015.04.002. Epub 2015 May 13. PMID 25979776